CLINICAL TRIAL: NCT00313937
Title: Single Centre, Open, Controlled, Randomised (1:1), Parallel Group: Insulin Glargine vs. NPH: FPG (Fasting Plasma Glucose) in Patients With DM Type 1 Who Skip the Morning Meal During Treatment With MDI (Multiple Daily Injection) Basal/Bolus Insulin
Brief Title: SAM - Skip a Meal - Insulin Glargine, Diabetes Mellitus Type 1
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Heinz Riederer / Medical Director, Sanofi-aventis Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HOE901_4028
Record Dates: First submitted 2006-04-11; First posted 2006-04-12 (Estimated); Last update posted 2009-12-07 (Estimated); Status verified 2009-12

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin Glargine

INTERVENTIONS:
Drug: Insulin glargine

SUMMARY:
Primary objective:

To compare metabolic control as measured by Blood Glucose (BG) upon arising from bed (7:00 am - 12:00 pm) in type 1 Diabetes mellitus patients who skip the morning meal during treatment with MDI basal/bolus insulin: Difference of change of blood glucose between 7:00 am and 11:00 am between patients on Insulin glargine and NPH insulin.

Secondary objective:

To perform an evaluation between the two patient groups for BG (10:00 pm and 12:00 pm) as well as for serum insulin, free fatty acid levels and β-hydroxybutyrate (7:00 am - 12:00 pm).

ELIGIBILITY:
Inclusion Criteria:

Patients with type 1 Diabetes mellitus who have been treated with MDI (Multiple Daily Injection) basal/bolus insulin, regular insulin/short acting insulin analogue + NPH insulin on a stable dose (no change more than 10 %) for at least 4 weeks prior to study entry, who have an HBA1c smaller/equal 9 % (measured at visit 1) and a BMI smaller/equal 35 kg/m2. In addition, patients must have a FBG value at day 1 before skipping meal (6:00 am - 07:00 am) between 90 - 120 mg/dl (5.0 - 6.5 mmol/l).

Exclusion Criteria:

* Breast-feeding
* History of hypersensitivity to the study medication or to drugs with similar chemical structures
* Likelihood of requiring treatment during the study period with drugs not permitted by the study protocol
* Treatment with any investigational drug in the last 30 days before study entry
* Clinically relevant cardiovascular, hepatic, neurological, endocrine, or other major systemic disease making implementation of the protocol or interpretation of the study results difficult
* History of drug or alcohol abuse

No subjects who have previously been treated with Insulin glargine will be enrolled in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2001-11; Primary Completion 2004-06 (Actual)

PRIMARY OUTCOMES:
Difference of change of blood glucose between patients on Insulin glargine and NPH insulin. | between 7:00 am and 11:00 am

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Landgraf, Dr., Study Director — Sanofi
Locations (1):
- Sanofi-Aventis, Berlin, Germany